CLINICAL TRIAL: NCT00857025
Title: A Phase I Study of MM-10-001 In Advanced Non Small Lung Cancer
Brief Title: Beta-Glucan in Treating Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07243; P30CA033572 (NIH); CHNMC-07243; CDR0000634737 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (beta-glucan MM-10-001) (Experimental): Patients receive oral beta-glucan MM-10-001 once or twice daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: beta-glucan MM-10-001; Other: flow cytometry; Other: laboratory biomarker analysis; Other: questionnaire administration

INTERVENTIONS:
Biological: beta-glucan MM-10-001 — Dose escalation with six patients treated at each of the following oral dosages: 2.5, 5.0, 7.5, 10, 15, 20, 30, 40, 50, and 80 mg/day
Other: flow cytometry — Performed on blood samples collected within 14 days prior to study treatment and at week 1, week 5, week 9, week 13 and every 4 weeks until the end of study treatment.
Other: laboratory biomarker analysis — Performed on blood samples collected within 14 days prior to study treatment and at week 1, week 5, week 9, week 13 and at the end of study treatment.
Other: questionnaire administration — Assessment pre-study and week 5, week 9, week 13 and at off study.

SUMMARY:
RATIONALE: Biological therapies, such as beta-glucan, may stimulate the immune system in different ways and stop tumor cells from growing.

PURPOSE: This phase I trial is studying the side effects and best dose of beta-glucan in treating patients with locally advanced or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the feasibility and toxicity of therapy with beta-glucan MM-10-001 in patients with locally advanced or metastatic non-small cell lung cancer for which standard curative or palliative measures do not exist or are no longer effective.

Secondary

* To explore analysis of the effect of beta-glucan MM-10-001 on the innate immune compartment, in particular natural killer cell activation and effector status.
* To perform correlatives (cytokine profiling) that will explore the effects of beta-glucan MM-10-001 on the cytokine profile of these patients.
* To document all clinical responses of these patients after treatment with beta-glucan MM-10-001.
* To explore potential beta-glucan MM-10-001 dose effects on the patient-reported functional status.

OUTLINE: Patients receive oral beta-glucan MM-10-001 once or twice daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for correlative studies. Samples are analyzed for natural killer cell activation and effector status and cytokine profiling by flow cytometry.

Patient-reported functional status is assessed at baseline and periodically during treatment by QOL-FACT-L questionnaire.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed non-small cell lung cancer

  * Locally advanced or metastatic disease for which standard curative or palliative measures do not exist or are no longer effective
  * Unresectable disease
* No active or symptomatic brain metastases unless they were previously treated by radiotherapy or surgery, stabilized, AND off steroid therapy for ≥ 4 weeks

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 50-100% OR ECOG PS 0-2
* Life expectancy > 3 months
* WBC > 2,000/mm³
* Absolute neutrophil count > 1,000/mm³
* Platelet count > 50,000/mm³
* Total bilirubin < 1.5 times upper limit of normal (ULN)
* AST and ALT < 2.5 times ULN
* Serum creatinine < 2.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must be able to swallow enteral medications (patients with feeding tubes are eligible)
* No condition or disease that affects gastrointestinal (GI) function or impairs the ability to take oral medications including any of the following:

  * GI tract disease
  * No intractable nausea or vomiting
  * Malabsorption syndrome
  * Requirement for IV alimentation
  * Prior surgical procedures effecting absorption
  * Uncontrolled inflammatory GI disease (e.g., Crohn disease, ulcerative colitis)
* No concurrent condition requiring the use of systemic or topical steroids or the use of immunosuppressive agents
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to beta-glucan MM-10-001
* No uncontrolled concurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) or radiotherapy and recovered

  * Concurrent palliative radiotherapy for symptoms control allowed
* At least 2 weeks since prior corticosteroids and no concurrent systemic or topical steroids
* At least 7 days since prior antioxidant supplements (vitamin C and E)
* No other concurrent investigational agents

  * Bisphosphonate therapy (e.g., pamidronate or zoledronate) allowed
* No concurrent over-the-counter or dietary supplement containing beta-glucan (e.g., mushroom extracts, "lentinan" products, dried mushrooms) or other mushroom-derived powders, liquids, capsules, gels, or any other dosage form
* No concurrent use of immunosuppressive agents (e.g., cyclosporine and its analog)
* No concurrent darbepoetin alfa or epoetin alfa
* No concurrent colony-stimulating factors
* No concurrent antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11-21 (Actual); Primary Completion 2010-11-24 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Safety | 28 days after therapy begins
Maximum-tolerated dose | 28 days after therapy begins
Toxicity as assessed by NCI CTCAE v3.0 | 28 days after therapy begins

SECONDARY OUTCOMES:
Beta-glucan MM-10-001 activity as assessed by changes in natural killer cell activation and functional activity, cytokine profiling, and clinical benefit | 13 weeks after start of study treatment
Patient-reported functional status | 13 weeks after start of study treatment
Survival | 1 year after start of study
Progression-free survival | 1 year after start of study

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Koczywas, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States